CLINICAL TRIAL: NCT06076876
Title: Prevalence and Risk Factors of Anxiety and Depression in Two Populations of Policemen During the Health Crisis Linked to COVID-19
Brief Title: Prevalence and Risk Factors of Anxiety and Depression Among Policemen During the Health Crisis Linked to COVID-19
Acronym: Covid19-Police
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8960
Record Dates: First submitted 2023-10-10; First posted 2023-10-11 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; Anxiety Syndrome; Depression Syndrome; Policemen
Keywords: Covid-19; Anxiety Syndrome; Depression Syndrome; Covid crisis; Police officers
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, there is little international data on depression and anxiety among police officers apart from studies carried out after an attack or natural disaster. At the national level, no mental health data exists for police officers, apart from those from the Paris attacks, and the work of investigators after the Strasbourg attack (article in press).

During the covid crisis, in Alsace, the police, like the rest of the population, took the full brunt of the pandemic. The police, however, are part of essential professions and have not been confined, but on the contrary, have remained in contact with the population, in particular to carry out traffic controls. Studies published to date show varying mental health outcomes for essential occupations during the pandemic.

The investigators hypothesize that the police officers had a feeling of being more exposed and that their mental health could be affected. For this it was decided to compare two populations of departments of similar size, but with different exposure to the pandemic: Bas Rhin and Hérault French departments

ELIGIBILITY:
Inclusion Criteria:

* Any major agent in office in June 2020 of the national police of the Bas Rhin department, and Hérault
* Supported between June and September 2020
* Subject not opposing, after information, the reuse of their data for the purposes of this research

Exclusion Criteria:

* Subject having expressed his opposition to his data being reused for study purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: National police officer in office in June 2020 in the departments of Bas Rhin and Hérault.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of depression and anxiety among policemen from two regions differently exposed to COVID 19 | 6 months after the covid crisis

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pathologie Professionnelle - Médecine du Travail - CHU de Strasbourg - France, Strasbourg, France